CLINICAL TRIAL: NCT04384965
Title: A Novel and Practical Accelerated Intermittent Theta Burst Protocol as a Substitute for Depressed Patients Needing Electroconvulsive Therapy During the COVID-19 Pandemic
Brief Title: Accelerated iTBS for Depressed Patients During the COVID-19 Pandemic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Principal Investigator, Daniel Blumberger, Medical Head and Co-Director, Temerty Centre for Therapeutic Brain Intervention, Centre for Addiction and Mental Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 059/2020
Record Dates: First submitted 2020-05-08; First posted 2020-05-12 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Major Depressive Disorder
Keywords: depression; transcranial magnetic stimulation; treatment resistance; theta burst stimulation
MeSH Terms: conditions — Depressive Disorder, Major; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Accelerated iTBS (Experimental): In the acute treatment phase, treatment will occur 8 times daily (50 min pause between treatments) on weekdays, until symptom remission is achieved (HRSD-24 score < to 10) or a maximum of 10 working days of daily treatment. In the tapering phase, treatments will be reduced to 2 treatment days per week for 2 weeks and then 1 treatment day per week for 2 weeks (4 weeks total). Patients will then enter the symptom-based relapse prevention phase including virtual check-in with study staff and a treatment schedule based on symptom level according to a modified relapse prevention algorithm that has been developed to prevent relapse after a successful course of ECT (known as the STABLE algorithm). The relapse prevention phase will last a maximum of 6 months.
  Interventions: Device: MagPro X100 Stimulator, B70 Fluid-Cooled Coil

INTERVENTIONS:
Device: MagPro X100 Stimulator, B70 Fluid-Cooled Coil — Treatment will occur 8 times per treatment day (50 min pause between treatments). Each treatment session will consist of a single iTBS treatment, delivering 600 pulses of iTBS (bursts of 3 pulses at 50 Hz, bursts repeated at 5 Hz, with a duty cycle of 2 seconds on, 8 seconds off, over 60 cycles / ~3 minutes) at a target of 110% of the subject's resting MT.

SUMMARY:
The current study aims to assess the feasibility, acceptance and clinical outcomes of a practical high-dose aiTBS protocol, including tapering treatments and symptom-based relapse prevention treatments, in patients with unipolar depression previously responsive to ECT and patients needing urgent treatment due to symptom severity during the COVID-19 pandemic.

ELIGIBILITY:
Inclusion Criteria:

* Have unipolar depressive episode based on the MINI with or without psychotic symptoms
* Have previous response to ECT or high symptom severity warranting acute ECT in the opinion of a consultant brain stimulation psychiatrist
* Are over the age of 18
* Pass the TMS adult safety screening (TASS) questionnaire
* Are voluntary and competent to consent to treatment

Exclusion Criteria:

* Have a Mini-International Neuropsychiatric Interview (MINI) confirmed diagnosis of substance dependence or abuse within the last 1 month
* Have a concomitant major unstable medical illness, cardiac pacemaker or implanted medication pump
* Have a lifetime Mini-International Neuropsychiatric Interview (MINI) diagnosis of bipolar I or II disorder, schizophrenia, schizoaffective disorder, schizophreniform disorder, delusional disorder
* Have any significant neurological disorder or insult including, but not limited to: any condition likely to be associated with increased intracranial pressure, space occupying brain lesion, any history of seizure except those therapeutically induced by ECT or a febrile seizure of infancy or single seizure related to a known drug related event, cerebral aneurysm, or significant head trauma with loss of consciousness for greater than 5 minutes
* have an intracranial implant (e.g., aneurysm clips, shunts, stimulators, cochlear implants, or electrodes) or any other metal object within or near the head, excluding the mouth, that cannot be safely removed
* currently take more than lorazepam 2 mg daily (or equivalent) or any dose of an anticonvulsant due to the potential to limit rTMS efficacy
* Lack of response to accelerated course of iTBS or rTMS in the past

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2020-05-12 (Actual); Primary Completion 2022-05-18 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
Proportion achieving remission on Hamilton Rating Scale for Depresion 24-it (HRSD-24) | Up to 10 days (From screening/baseline to end of the acute treatment)
  Less than or equal to 10

SECONDARY OUTCOMES:
Change in HRSD-24 | Up to 10 days (From screening/baseline to end of the acute treatment)
  changes in scores
Response on HRSD-24 | Up to 10 days (From screening/baseline to end of the acute treatment)
  50% Reduction in score
Remission on Patient Health Questionnaire (PHQ-9) | Up to 10 days (From screening/baseline to end of the acute treatment)
  Less than or equal to 4
Response on PHQ-9 | Up to 10 days (From screening/baseline to end of the acute treatment)
  50% Reduction in score
Change in PHQ-9 | Up to 10 days (From screening/baseline to end of the acute treatment)
  changes in scores
Remission on General Anxiety Disorder 7 item (GAD-7) | Up to 10 days (From screening/baseline to end of the acute treatment)
  Less than or equal to 4
Response on GAD-7 | Up to 10 days (From screening/baseline to end of the acute treatment)
  50% Reduction in score
Change in GAD-7 | Up to 10 days (From screening/baseline to end of the acute treatment)
  changes in scores
Remission on Beck Depression Inventory (BDI-II) | Up to 10 days (From screening/baseline to end of the acute treatment)
  Less than or equal to 12
Response on BDI-II | Up to 10 days (From screening/baseline to end of the acute treatment)
  50% Reduction in Score
Change on BDI-II | Up to 10 days (From screening/baseline to end of the acute treatment)
  changes in scores
Remission on Beck Scale for Suicidal Ideation (SSI) | Up to 10 days (From screening/baseline to end of the acute treatment)
  Score of 0
Change on SSI | Up to 10 days (From screening/baseline to end of the acute treatment)
  changes in scores
Change in WHO Disability Assessment Schedule (WHODAS) | Up to 10 days (From screening/baseline to end of the acute treatment)
  changes in scores
Proportion of Patients Maintaining Response During Relapse Prevention | 24 weeks (Tapering and Relapse prevention phase)
  Includes number of treatment days needed and number going on to receive ECT

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Blumberger, MD, Principal Investigator — CAMH
Locations (1):
- CAMH, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Goodman MS, Trevizol AP, Konstantinou GN, Boivin-Lafleur D, Brender R, Downar J, Kaster TS, Knyahnytska Y, Vila-Rodriguez F, Voineskos D, Daskalakis ZJ, Blumberger DM. Extended course accelerated intermittent theta burst stimulation as a substitute for depressed patients needing electroconvulsive therapy. Neuropsychopharmacology. 2025 Mar;50(4):685-694. doi: 10.1038/s41386-024-02007-w. Epub 2024 Oct 23. PMID 39443721